CLINICAL TRIAL: NCT03826173
Title: Physical Activity Promotion Based on Positive Psychology: Development and Piloting of a Novel Intervention Approach
Brief Title: Positive Psychology for Physical Activity Promotion
Acronym: PPPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21CA224609-01A1 (NIH); 1R21CA224609-01A1 (NIH)
Record Dates: First submitted 2018-09-18; First posted 2019-02-01 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Physical Activity
Keywords: Positive Psychology; Affect
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology (Experimental): On a weekly basis, participants will engage in group-based intervention sessions that focus on personal strengths and the value of positive emotions and cognitions. Participants will receive daily text-messages addressing the content introduced during group sessions.
  Interventions: Behavioral: PPPA
- Physical Activity Promotion (Active Comparator): On a weekly basis, participants will engage in group-based intervention sessions that focus on the standard physical activity promotion components of the PPPA condition. Participants will receive daily text-messages addressing the content introduced during group sessions.
  Interventions: Behavioral: PA

INTERVENTIONS:
Behavioral: PPPA — The intervention will focus on a) health benefits of PA, b) individualized PA intensity prescriptions and instruction on gauging PA intensity, c) goal-setting and self-monitoring, and d) tips on overcoming barriers to PA. Participants will be instructed to target 30-60 min/day 5 days/week of MVPA consistent with national guidelines. PA content will be concentrated in sessions 1 and 2, but content on goal-setting, self-monitoring, and overcoming barriers will continue throughout the 6-week period. The intervention includes activities that focus on identifying each individual's strengths, identifying/savoring positive experiences, engaging in constructive conversation, expressing gratitude, and strategies to maintain increased positive affect after the intervention has completed.
  Arms: Positive Psychology
Behavioral: PA — The intervention will focus on (a) health benefits of PA, (b) individualized PA intensity prescriptions and instruction on how to gauge PA intensity, (c) goal-setting and self-monitoring, and (d) tips on overcoming barriers to PA, including time-management. Participants will be instructed to target 30-60 min/day 5 days/week of MVPA consistent with national guidelines. PA content will be concentrated in sessions 1 and 2, but content on goal-setting, self-monitoring, and overcoming barriers will continue throughout the 6-week period.
  Arms: Physical Activity Promotion

SUMMARY:
This study is for physically inactive adults. Participants will be enrolled in the Positive Psychology and Physical Activity intervention designed to help them overcome barriers to physical activity, based on the principals of positive psychology.

This will involve six weekly one-hour group-based sessions at a local YMCA with a trained group leader. In addition to the in-person sessions, there will be text messages sent to participants about physical activity that include positive psychology content.

DETAILED DESCRIPTION:
The investigators propose to conduct a pilot study to test feasibility and proof-of-concept for a positive psychology intervention program to promote exercise among low-active overweight and obese adults. The program will be (a) a 6-week, group-based intervention, (b) delivered at local YMCAs, and (c) supplemented with text messaging. In an additive design, participants will be randomized in a 2:1 ratio to PPPA (n = 40) versus a control intervention (n = 20) including only the standard PA promotion components of the PPPA intervention (i.e., PA education, self-monitoring, and goal-setting), with equal frequency of staff contact and text message delivery. All participants will be followed for 3 months, and will receive a 3-month YMCA membership to equate access to PA facilities. As a secondary aim the investigators will examine effect sizes for PPPA versus the standard PA intervention on putative mediators that may underlie the efficacy of PPPA in improving PA outcomes, including positive and negative affect, optimism, happiness, life satisfaction, social support for PA, and PA enjoyment. The proposed research will set the stage for an RCT to test a novel PA promotion intervention that can be readily disseminated.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary or low-active, (defined as < 60 min/week of structured physical activity)
* Able to receive and respond to a text message at the time of screening

Exclusion Criteria:

* History of coronary artery disease
* History of stroke
* History of uncontrolled hypertension
* History of asthma
* History of chronic obstructive pulmonary disease (COPD)
* History of diabetes
* History of osteoarthritis or orthopedic problems that limit physical activity
* BMI greater than 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Williams, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with interested parties after all of the initial study analyses and outcomes have been published.
Time Frame: Data will be made available 1 year after the completion of the study.
Access Criteria: All data access requests will be reviewed by a panel prior to acceptance.

RESULTS

PARTICIPANT FLOW:
Groups:
- Positive Psychology Phase 1; Positive Psychology Phase 2: On a weekly basis, participants will engage in group-based intervention sessions that focus on personal strengths and the value of positive emotions and cognitions. Participants will receive daily text-messages addressing the content introduced during group sessions.
  PPPA: The intervention will focus on a) health benefits of PA, b) individualized PA intensity prescriptions and instruction on gauging PA intensity, c) goal-setting and self-monitoring, and d) tips on overcoming barriers to PA. Participants will be instructed to target 30-60 min/day 5 days/week of MVPA consistent with national guidelines. PA content will be concentrated in sessions 1 and 2, but content on goal-setting, self-monitoring, and overcoming barriers will continue throughout the 6-week period. The intervention includes activities that focus on identifying each individual's strengths, identifying/savoring positive experiences, engaging in constructive conversation, expressing gratitude, and strategies to maintain increased positive affect after the intervention has completed.
Period: Overall Study
Arm/Group | Positive Psychology Phase 1 | Positive Psychology Phase 2 | Physical Activity Promotion
Started | 13 | 30 | 11
Completed | 12 | 27 | 6 (Treatment was cut short by COVID-19)
Not Completed | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Psychology Phase 1 | Positive Psychology Phase 2 | Physical Activity Promotion | Total
Number analyzed (Participants) | 13 | 30 | 11 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (12.8) | 40.1 (14.5) | 37.3 (15.2) | 40.9 (14.3)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender: 1=male, 2=female, 3=non-binary/third gender, 4=prefer to self-describe, 5=prefer not to say
  Participants
    Male | 1 | 13 | 2 | 16
    Female | 12 | 16 | 9 | 37
    Prefer not to say | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 3 | 13
  Not Hispanic or Latino | 9 | 23 | 8 | 40
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 1 | 7
  White | 10 | 18 | 6 | 34
  More than one race | 1 | 1 | 2 | 4
  Unknown or Not Reported | 1 | 4 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Moderate-to-Vigorous Minutes of Physical Activity Per Week
Description: Change in Moderate-to-Vigorous Minutes of Physical Activity Per Week [Time Frame: Measured at baseline, mid-treatment (week 4), and post-treatment (week 7).]
Time Frame: Measured at baseline, mid-treatment (week 4), and post-treatment (week 7).
Population: Reporting of raw means. This is a feasibility study. It lacks adequate power for inferential analysis.
Measure: Mean (Standard Deviation); unit: Minutes of physical activity
Arm/Group | Positive Psychology Phase 1 | Positive Psychology Phase 2 | Physical Activity Promotion
Number analyzed (Participants) | 13 | 30 | 11
Minutes of physical activity
  Baseline | 27.4 (51.8) | 83.0 (105.1) | 88.4 (77.6)
  Mid-treatment: number analyzed (Participants) | 12 | 30 | 6
  Mid-treatment | 54.5 (50.2) | 95.1 (84.6) | 140.7 (97.9)
  Post-treatment: number analyzed (Participants) | 12 | 27 | 6
  Post-treatment | 21.9 (29.7) | 125.4 (107.2) | 61.0 (61.2)

2. Secondary Outcome: Change in Positive and Negative Affect
Description: The Positive and Negative Affect Scale measures changes in positive and negative affect. Both positive and negative affect sub-scales will be scored (scores range from 10 to 50 for each individual sub-scale), with higher scores on the positive affect scale and lower scores on the negative affect scale indicating a better outcome.
Time Frame: Survey will be administered at baseline, week 4 (mid-treatment), week 7 (post-treatment), and week 10 (one-month follow-up).
Reporting Status: Not Posted

3. Secondary Outcome: Change in Optimism
Description: Life Orientation Test- Revised measures trait optimism. Scores range from 10 to 50, with higher scores reflecting greater optimism. Higher scores will reflect better outcomes of the intervention.
Time Frame: as for outcome 2
Reporting Status: Not Posted

4. Secondary Outcome: Change in Subjective Happiness
Description: Measure of subjective happiness. Scores range from 4 to 28, with higher scores reflecting greater subjective happiness. Higher scores will reflect better outcomes of the intervention.
Time Frame: Survey will be administered at baseline, week 4, week 7, and week 10.
Reporting Status: Not Posted

5. Secondary Outcome: Change in Satisfaction With Life
Description: Measures subjective well-being. Scores range from 5 to 35, with higher scores reflecting greater satisfaction with life and subjective well-being. Higher scores will reflect better outcomes of the intervention.
Time Frame: as for outcome 2
Reporting Status: Not Posted

6. Secondary Outcome: Change in Social Support for Exercise
Description: Measures perceived social support for regular exercise. Scores range from 13 to 65, with higher scores reflecting greater social support. Will be assessed as a putative mediator.
Time Frame: as for outcome 2
Reporting Status: Not Posted

7. Secondary Outcome: Change in Physical Activity Enjoyment
Description: Measures enjoyment of physical activity. Scores range from 18 to 126, with higher scores reflecting greater enjoyment. Will be assessed as a putative mediator.
Time Frame: as for outcome 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Six weeks per participant
Arm/Group | Positive Psychology Phase 1 | Positive Psychology Phase 2 | Physical Activity Promotion
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/30 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/30 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/30 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT03826173/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT03826173/ICF_001.pdf